CLINICAL TRIAL: NCT05721027
Title: Ibuprofen With or Without Dexamethasone for Acute Radicular Low Back Pain.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-14723
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Radiculopathy, Lumbosacral Region; Back Pain With Radiation; Low Back Pain
Keywords: ibuprofen; dexamethasone; radiculopathy; low back pain; back pain with radiation
MeSH Terms: conditions — Radiculopathy; Back Pain; Low Back Pain | interventions — Ibuprofen; Dexamethasone; Early Intervention, Educational

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ibuprofen + dexamethasone + educational intervention (Experimental): Ibuprofen 400 mg PO every 8 hours as needed for 7 days + dexamethasone 16 mg PO for day 1 and day 2. Research personnel will provide each participant with a 15-minute educational intervention.
  Interventions: Drug: Ibuprofen 400 mg; Drug: Dexamethasone Oral; Behavioral: Educational Intervention
- Ibuprofen + placebo + educational intervention (Placebo Comparator): Ibuprofen 400 mg PO every 8 hours as needed for 7 days + placebo PO for day 1 and day 2. Research personnel will provide each participant with a 15-minute educational intervention.
  Interventions: Drug: Ibuprofen 400 mg; Behavioral: Educational Intervention

INTERVENTIONS:
Drug: Ibuprofen 400 mg — Ibuprofen 400 mg PO every 8 hours as needed for 7 days
Drug: Dexamethasone Oral — Dexamethasone 16 mg PO during ED visit and next day
  Arms: Ibuprofen + dexamethasone + educational intervention
Behavioral: Educational Intervention — Research personnel will provide each patient with a 15-minute educational intervention. This will be based on National Institute of Arthritis and Musculoskeletal and Skin Diseases Handout on Health: Back Pain information

SUMMARY:
This will be a placebo controlled, randomized, double-blind, comparative effectiveness study, in which we patients are enrolled during an emergency department (ED) visit for acute radicular low back pain (LBP) and followed by telephone two and seven days later. Patients will be randomized to receive an oral dose of dexamethasone for 2 consecutive days or placebo during an ED visit for acute radicular LBP. Every patient will receive a 7 day supply of ibuprofen and a low back pain education session.

ELIGIBILITY:
Inclusion Criteria:

* Present to ED primarily for management of acute radicular LBP, defined as pain or paresthesia originating from the lower back and radiating to the buttock and or leg in a radicular pattern. Some patients may not have prominent LBP but a radicular symptom--we will include these patients as well.
* Patient is to be discharged home.
* Age 18-70 Enrollment will be limited to adults <70 years because of the increased risk of adverse medication effects in older adults.
* Pain duration <2 week
* Prior to the acute attack of radicular LBP, back pain cannot occur more frequently than half of the days in the last 3 months. Patients with more frequent back pain/sciatica are at increased risk of poor pain and functional outcomes.10
* Non-traumatic cause of pain: no substantial and direct trauma to the back within the previous month
* Functionally impairing radicular LBP: A baseline score of > 5 on the Roland-Morris Disability Questionnaire

Exclusion Criteria:

* Not available for follow-up
* Pregnant
* Chronic pain syndrome defined as use of any analgesic medication on a daily or near-daily basis
* Allergic to or intolerant of investigational medications
* Chronic steroid use
* Contra-indications to investigational medications: 1) known peptic ulcer disease, chronic dyspepsia, or history of gastrointestinal bleed 2) Severe heart failure (NYHA 2 or worse) 3) Chronic kidney disease (GFR <60ml/min) 4) Current use of anti-coagulants 5) cirrhosis (Child Pugh A or worse) or hepatitis (transaminases 2x the upper limit of normal)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in Roland Morris Disability Questionnaire (RMDQ) score | 2 days (48 hours)
  The change in RMDQ will be evaluated using the 24-item Roland Morris Low Back Pain Disability Questionnaire. The RMDQ is a 24-item patient-reported outcome measure that inquires about pain-related disability resulting from LBP. Items are scored 0 if left blank or 1 if endorsed, for a total RMDQ score ranging from 0 to 24. Higher scores represent higher levels of pain-related disability. The change will be calculated as a difference between the baseline ED visit and the two day follow-up visit (Roland-Morris baseline - Roland-Morris day 2)

SECONDARY OUTCOMES:
Worst Radicular LBP | 2 days and 7 days after ED discharge
  Worst Radicular LBP pain incurred over the previous 24 hours will be assessed at 2 days and 7 days after ED discharge using a four point ordinal scale: Severe, Moderate, Mild, or None
Frequency of Radicular LBP | 2 days and 7 days after ED discharge
  Frequency of Radicular LBP is evaluated at 2 days and 7 days after ED discharge based on a five point Likert scale: Not at all, Rarely, Sometimes, Usually, and Always
Analgesic or LBP medication within the previous 24 hours | 2 days and 7 days after ED discharge
  Administration of any analgesic or LBP medication (Yes or No) within the previous 24 hours will be assessed at 2 days and 7 days after ED discharge
Absolute Roland Morris Disability Questionnaire (RMDQ) score | 2 days and 7 days after ED discharge
  The Absolute RMDQ score will be tabulated at 2 days and 7 days after ED discharge. The RMDQ is a 24-item patient-reported outcome measure that inquires about pain-related disability resulting from LBP. Items are scored 0 if left blank or 1 if endorsed, for a total RMDQ score ranging from 0 to 24. Higher scores represent higher levels of pain-related disability
Return to all usual activities | 2 days and 7 days after ED discharge
  The patient will be evaluated for the ability to return to all usual activities at 2 days and 7 days after ED discharge based on a binary (Yes/No) response
Number of visits to any healthcare provider | 2 days and 7 days after ED discharge
  The number of aggregate visits to any healthcare provider will be tabulated at 2 days and 7 days after ED discharge
Satisfaction with Treatment | 2 days and 7 days after ED discharge
  Satisfaction with treatment will be evaluated based on a binary (Yes/No) response at 2 days and 7 days after ED discharge

CONTACTS AND LOCATIONS:
Overall Officials: Eddie Irizarry, MD, Principal Investigator — Montefiore Medical Center
Locations (2):
- United States (2):
  - Albert Einstein College of Medicine/Montefiore Medical Center - Weiler ED, The Bronx, New York
  - Montefiore Medical Center - Moses ED, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No
No plan to share

REFERENCES:
- See also: National Institute of Arthritis and Musculoskeletal and Skin Diseases Handout on Health: Back Pain information — https://www.niams.nih.gov/health-topics/back-pain